CLINICAL TRIAL: NCT04731948
Title: A Dose-finding Randomized Trial of Vitamin B12 Supplementation: Biomarker Responses and Implications for Dietary Recommendations.
Brief Title: Vitamin B12 Biomarker Responses to Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: University of Dublin, Trinity College (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UUREC 04/38
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Vitamin B12; Serum holotranscobalamin; Serum total vitamin B12; Dietary recommendations; Plasma methylmalonic acid; Plasma homocysteine
MeSH Terms: interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: A double-blind randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Folic Acid + Placebo (Placebo Comparator): 400µg Folic Acid per day for 16 weeks after a pre-treatment phase with 400µg FA per day for 11 weeks
  Interventions: Dietary Supplement: Folic Acid
- Folic Acid + Vitamin B12 Dose 1 (Active Comparator): 400µg Folic Acid + 2 µg Vitamin B12 per day for 16 weeks after a pre-treatment phase with 400µg FA per day for 11 weeks
  Interventions: Dietary Supplement: Folic Acid; Dietary Supplement: 2 µg Vitamin B12
- Folic Acid + Vitamin B12 Dose 2 (Active Comparator): 400µg Folic Acid + 10 µg Vitamin B12 per day for 16 weeks after a pre-treatment phase with 400µg FA per day for 11 weeks
  Interventions: Dietary Supplement: Folic Acid; Dietary Supplement: 10 µg Vitamin B12
- Folic Acid + Vitamin B12 Dose 3 (Active Comparator): 400µg Folic Acid + 50 µg Vitamin B12 per day for 16 weeks after a pre-treatment phase with 400µg FA per day for 11 weeks
  Interventions: Dietary Supplement: Folic Acid; Dietary Supplement: 50 µg Vitamin B12

INTERVENTIONS:
Dietary Supplement: Folic Acid — 400µg Folic Acid per day for 16 weeks
Dietary Supplement: 2 µg Vitamin B12 — 2 µg Vitamin B12 per day for 16 weeks
  Arms: Folic Acid + Vitamin B12 Dose 1
Dietary Supplement: 10 µg Vitamin B12 — 10 µg Vitamin B12 per day for 16 weeks
  Arms: Folic Acid + Vitamin B12 Dose 2
Dietary Supplement: 50 µg Vitamin B12 — 50 µg Vitamin B12 per day for 16 weeks
  Arms: Folic Acid + Vitamin B12 Dose 3

SUMMARY:
The aim of the study is to investigate the response of recognized biomarkers of vitamin B12 status to intervention with supplemental vitamin B12 at doses within and beyond the range of typical dietary intakes in younger and older adults.

Study design: A double-blind randomized controlled trial in healthy adults aged 18 years and over will be conducted. Apparently healthy individuals will be recruited from the staff and student population at Ulster University, Coleraine, and the surrounding local community. Those interested in the study will provide informed consent. Individuals suffering from chronic conditions, those taking medications interfering with folate or vitamin B12 metabolism or B vitamin supplements, and women who are pregnant will be excluded from participation. Potential participants will provide a non-fasting blood sample and those with plasma creatinine concentration > 130 µmol/L, those with hypochlorhydria (diagnosed serologically by pepsinogen I to Pepsinogen II ratio < 3) and those with the 677C→T polymorphism in the methylenetetrahydrofolate reductase (MTHFR) gene will also be excluded from the study. In addition, participants aged 60 years and over who score <25 on the Folstein's Mini-Mental State Examination (a cognitive function screening test) will be excluded to reduce the risk of including participants with impaired cognitive function and thus reduced ability to comply with the study requirements, including compliance with the intervention trial and recall of food intake.

All eligible participants will undergo a pre-treatment phase with 400 µg/day folic acid (FA) for 11 weeks. At the end of this phase, participants will provide a non-fasting blood sample (baseline sample) and will be stratified within each age category (<60 years and ≥60 years) according to their homocysteine concentrations and subsequently randomized from each stratum (in a 1:1:1:1 allocation ratio) to one of the four treatments for 16 weeks: 400 µg/day FA + placebo, 400 µg/day FA + 2 µg/day vitamin B12, 400 µg/day FA + 10 µg/day vitamin B12 or 400 µg/day FA + 50 µg/day vitamin B12. A non-fasting blood sample will be collected at the end of the intervention. Biomarkers of vitamin B12 and folate will be measured in blood samples collected at baseline and post-intervention. The intervention will be conducted on a staggered basis and both study participants and researchers will be blinded to the treatment allocations. Dietary intake of participants will be assessed using a four-day food diary based on 2 weekday and 2 weekend day intakes in combination with a food frequency questionnaire particularly focused on intakes of foods fortified with vitamin B12 and FA.

DETAILED DESCRIPTION:
Detailed Description:

The aim of this study is to investigate the response of recognized vitamin B12 biomarkers (serum total vitamin B12; serum holotranscobalamin; plasma methylmalonic acid; plasma homocysteine) to intervention with supplemental vitamin B12 at doses within and beyond the range of typical dietary intakes in younger and older adults.

The sample size will be estimated by using typical variances from published studies on plasma homocysteine responses to vitamin B12 supplementation in adults. The calculations are based on changes in plasma homocysteine, as it is considered a functional indicator of vitamin B12 status. The typical standard deviation of change will be set at 2µmol/L (Clarke et al. 1998; McKinley et al. 2002) with the minimal detectable difference being 1.5µmol/L at 80% power and a significance level of 5%. Calculations determined that 40 subjects would be required for each of the three treatment groups plus placebo in order to show significant differences in plasma homocysteine concentrations.

Participants will be recruited by posters, advertisement, emails and organized meetings to promote the study among staff and students at Ulster University, Coleraine, workplaces, social and sporting clubs and sheltered accommodation for older adults in the surrounding local community. Those interested in the study will receive a participant information sheet and further details about the study. A signed informed consent will be obtained from all who are willing to participate in the study. A screening questionnaire and a non-fasting blood sample will be taken to identify those eligible to take part in the study. Exclusion criteria will be: history of gastrointestinal, hepatic, renal, vascular or haematological diseases or diabetes; those taking medications that interfere with folate or vitamin B12 metabolism (e.g. methotrexate, proton pump inhibitor drugs); use of B vitamin supplements; pregnancy; plasma creatinine concentration > 130 µmol/L; those with hypochlorhydria (diagnosed serologically by pepsinogen I to Pepsinogen II ratio < 3); those individuals with the 677C→T polymorphism in the MTHFR gene and those aged 60 years and over who scored <25 on Folstein's Mini-Mental State Examination (a cognitive function screening test).

All eligible participants will undergo a pre-treatment phase with 400 µg/day folic acid (FA) for 11 weeks; the treatment with FA will continue until the end of the trial. At the end of the pre-treatment phase, participants will provide a non-fasting blood sample (baseline sample) and will be stratified within each age category (<60 years and ≥60 years) according to their homocysteine concentrations and subsequently randomized in a 1:1:1:1 allocation ratio to one of the four treatments for 16 weeks: 400 µg/day FA + placebo, 400 µg/day FA + 2 µg/day vitamin B12, 400 µg/day FA + 10 µg/day vitamin B12 or 400 µg/day FA + 50 µg/day vitamin B12. A non-fasting blood sample will be collected at the end of the intervention. Blood samples at baseline and post-intervention will be analyzed for biomarkers of folate and vitamin B12 status. In order to encourage maximal compliance, participants will be contacted regularly and provided with supplements in 7-day pillboxes every 4 weeks during the pre-treatment phase and the intervention, and will be asked to return the used pillboxes; the number of unused capsules will be recorded to monitor compliance. The intervention will be conducted on a staggered basis and both study participants and researchers will be blind to treatment allocations. Dietary intake of participants will be assessed using a four-day food diary (based on 2 weekday and 2 weekend day intakes) and a food frequency questionnaire regarding specific intake of foods fortified with vitamin B12 and FA.

Anthropometric measurements as height and weight for each participant will be taken by using portable approved scales.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 years and above who do not comply with the exclusion criteria

Exclusion Criteria:

* History of gastrointestinal, hepatic, renal, vascular or haematological diseases, or diabetes;
* Use of medication known to interfere with B12 metabolism (e.g. methotrexate, proton pump inhibitor drugs);
* Use of B vitamin supplements;
* Pregnancy;
* Plasma creatinine concentration > 130 µmol/L;
* Hypochlorhydria (diagnosed serologically by pepsinogen I to Pepsinogen II ratio < 3);
* Score of less than 25 on Folstein's Mini-Mental State Examination (a cognitive function screening test; for people aged 60 years and over);
* 677C→T polymorphism in the MTHFR gene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-10-01 (Actual); Primary Completion 2006-12-12 (Actual); Study Completion 2006-12-12 (Actual)

PRIMARY OUTCOMES:
Vitamin B12 biomarkers | Change between screening (before pre-treatment phase), baseline (after pre-treatment phase) and post-intervention (16 weeks)
  Serum vitamin B12 concentrations measured by a microbiological L. Leichmannii assay
Vitamin B12 biomarkers | Change between screening (before pre-treatment phase), baseline (after pre-treatment phase) and post-intervention (16 weeks)
  Serum holotranscobalamin concentrations measured by a AxSym based immunoassay
Vitamin B12 biomarkers | Change between screening (before pre-treatment phase), baseline (after pre-treatment phase) and post-intervention (16 weeks)
  Plasma methylmalonic acid concentrations measured by Gas Chromatography-Mass Spectrometry
Vitamin B12 biomarkers | Change between screening (before pre-treatment phase), baseline (after pre-treatment phase) and post-intervention (16 weeks)
  Plasma homocysteine concentrations measured by a fluorescence polarization immunoassay

SECONDARY OUTCOMES:
Folate status | Change between screening (before pre-treatment phase), baseline (after pre-treatment phase) and post-intervention (16 weeks)
  Serum and red blood cell folate concentrations measured by a microbiological L. casei assay;
MTHFR C677T polymorphism (rs1801133) | At screening (before pre-treatment phase)
  Determined by polymerase chain reaction amplification followed by Hin F1 restriction digestion enzyme
Serum Pepsinogen concentrations | At screening (before pre-treatment phase)
  Serum Pepsinogen I and pepsinogen II concentrations measured by ELISA kits
Plasma creatinine | At screening (before pre-treatment phase)
  Plasma creatinine assessed by a standard spectrophotometric
BMI | At baseline (after pre-treatment phase)
  Height (cm) and weight (kg) for the calculation of BMI
Cognition | At screening (before pre-treatment phase)
  Folstein's Mini-Mental State Examination for potential participants aged 60 years and over

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom